CLINICAL TRIAL: NCT01687972
Title: A Randomized Controlled Trial of Skin Closure at Cesarean Section: INSORB Absorbable Staples Versus Subcuticular Sutures
Brief Title: INSORB Versus Subcuticular Sutures at Cesarean Section
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00043795
Record Dates: First submitted 2012-09-09; First posted 2012-09-19 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-08

CONDITIONS: Cesarean Section; Pregnancy
Keywords: cesarean section; insorb staples; absorbable staples; transverse skin incision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sutures (Active Comparator)
  Interventions: Combination Product: Absorbable sutures
- Insorb Staples (Active Comparator)
  Interventions: Combination Product: Insorb absorbable staples

INTERVENTIONS:
Combination Product: Insorb absorbable staples — Placement of Insorb absorbable staples at cesarean section
  Arms: Insorb Staples
Combination Product: Absorbable sutures — placement of absorbable sutures at cesarean section
  Arms: Sutures

SUMMARY:
The proposed study is a randomized controlled trial with two arms. All patients admitted to Labor and Delivery at Johns Hopkins Hospital for delivery will be approached and offered entry into our study. Once the patient is enrolled, and if she undergoes a cesarean section, the patient will be randomized at time of cesarean section to receive skin closure by either the INSORB™ absorbable staples or subcuticular closure using Biosyn™ suture as is the standard practice. Both an observer scar assessment score (OSAS) and patient scar assessment score (PSAS) will be obtained during this visit. The patient will then be contacted by telephone by a study member 3 months after her surgery for a brief survey (same PSAS survey) assessing her satisfaction with the resulting scar.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial with two arms. All patients admitted to Labor and Delivery at Johns Hopkins Hospital for delivery will be approached and offered entry into our study during the routine consent process which includes consent for cesarean section that occurs with each patient. Once the patient is enrolled, and if she undergoes a cesarean section, the patient will be randomized at time of cesarean section to receive skin closure by either the INSORB™ absorbable staples or subcuticular closure using Biosyn™ suture as is the standard practice. The size of the suture (3-0 vs. 4-0) and type of needle used to sew is at the discretion of the surgeon. The indications for and performance of the cesarean section will remain standard care by the Obstetrical team and the patient's participation in this study will have no impact whatsoever on the obstetrical course of the patient. The only additional procedure that will be asked of the obstetrical team performing the cesarean section is to measure and close the subcutaneous tissue if the depth from the skin edge to the transversalis fascia is greater than 2cm as this has been shown to decrease subsequent seroma formation and wound disruption. The dressing will be standardized as follows: a folded abdominal (ABD) pad will be placed in a sterile fashion directly over the incision and foam tape will be applied to provide a "pressure dressing." The dressing will be removed on post-operative day #2.

The patient's postoperative course will remain unchanged and her discharge will be at the discretion of her obstetrical providers. On post-operative day #3, a picture of the incision will be taken with the patient's identifying number adjacent to the picture and the patient will be asked to complete a brief survey asking about post-operative pain and scars (see included PSAS survey). The patients will follow-up with her Obstetrician for her normal post-partum visit where another picture of the incision will be taken. Both an observer scar assessment score (OSAS) and patient scar assessment score (PSAS) will be obtained during this visit. The patient will then be contacted by telephone by a study member 3 months after her surgery for a brief survey (same PSAS survey) assessing her satisfaction with the resulting scar. At this point, the patient's participation in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* cesarean section via transverse skin incision informed consent

Exclusion Criteria:

* vertical skin incision

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Chelmow D, Rodriguez EJ, Sabatini MM. Suture closure of subcutaneous fat and wound disruption after cesarean delivery: a meta-analysis. Obstet Gynecol. 2004 May;103(5 Pt 1):974-80. doi: 10.1097/01.AOG.0000124807.76451.47. PMID 15121573
- [Background] Basha SL, Rochon ML, Quinones JN, Coassolo KM, Rust OA, Smulian JC. Randomized controlled trial of wound complication rates of subcuticular suture vs staples for skin closure at cesarean delivery. Am J Obstet Gynecol. 2010 Sep;203(3):285.e1-8. doi: 10.1016/j.ajog.2010.07.011. PMID 20816153
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924
- [Background] Gaertner I, Burkhardt T, Beinder E. Scar appearance of different skin and subcutaneous tissue closure techniques in caesarean section: a randomized study. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):29-33. doi: 10.1016/j.ejogrb.2007.07.003. Epub 2007 Sep 6. PMID 17825472
- [Background] Couto RC, Pedrosa TM, Nogueira JM, Gomes DL, Neto MF, Rezende NA. Post-discharge surveillance and infection rates in obstetric patients. Int J Gynaecol Obstet. 1998 Jun;61(3):227-31. doi: 10.1016/s0020-7292(98)00047-2. PMID 9688482
- [Background] Menacker F, Hamilton BE. Recent trends in cesarean delivery in the United States. NCHS Data Brief. 2010 Mar;(35):1-8. PMID 20334736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 187 were consented, and 88 were randomized to intervention versus placebo.
Period: Overall Study
Arm/Group | Sutures | Insorb Staples
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sutures | Insorb Staples | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Scale
Description: Visual Analog Score 0-10, with 0 being painless and 10 being the most severe
Time Frame: 3 months
Population: Data was not collected for all participants enrolled due to failure to follow-up post intervention.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sutures | Insorb Staples
Number analyzed (Participants) | 19 | 16
units on a scale | 2.375 [1 to 8] | 3.053 [0 to 10]

2. Primary Outcome: Patient Scar Assessment Scale (PSAS)
Description: assessed using the Objective scar scale score, score range 6-60 with 6 being the best score, representing normal skin and 60 being the worst score representing scar very different from the normal skin.
Time Frame: 6 weeks
Population: Data was unable to be collected from all participants randomized due to lack of follow-up post intervention.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sutures | Insorb Staples
Number analyzed (Participants) | 2 | 1
units on a scale | 20 [11 to 29] | 13 [13 to 13]

3. Primary Outcome: Closure Time
Description: Number of minutes taken to close post cesarean section
Time Frame: up to 20 minutes post intervention
Population: Data was not collected for all participants enrolled
Measure: Mean (Full Range); unit: minutes
Arm/Group | Sutures | Insorb Staples
Number analyzed (Participants) | 33 | 31
minutes | 4.161 [1 to 8] | 9.79 [1 to 16]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Sutures | Insorb Staples
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes